CLINICAL TRIAL: NCT03789539
Title: Reactogenicity, Safety and Immunogenicity of an Recombinant Universal Influenza Vaccine Uniflu in Healthy Volunteers From 18 to 60 Years Old
Brief Title: Reactogenicity, Safety and Immunogenicity of an Universal Influenza Vaccine Uniflu
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VA Pharma Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UIV-I-01/2017
Record Dates: First submitted 2018-12-24; First posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Safety Issues
Keywords: Safety; Reactogenicity; Universal Influenza Vaccine

STUDY DESIGN:
Intervention Model Description: Subjects will undergo screening procedures within 2-6 days prior to first vaccination which will include medical history, vital signs, physical examination and safety blood and urine lab tests.
  On the first treatment visit, eligible subjects will undergo pre-dose physical examination, ECG, vital signs, and a blood sample for circulating IgE. They will then receive an IM injection of either vaccine or placebo, according to the above treatment assignment, into the deltoid muscle preferably of non dominant arm. The subjects will remain under medical supervision for 72 hrs at which time they will be released from the Clinical research center.
  The second treatment will take place 21 days after the first vaccination. Procedures will be the same as that of Visit 1 Additional follow-up visits will take place at 4-7th,14th,24-27th and 42nd days. Blood and urine samples will be collected for safety.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LD Universal Influenza Vaccine Uniflu (Active Comparator): low dose of Uniflu vaccine 0.5 ml (20 mkg of recombinant protein HBc-4M2eh) administrated intramuscularly 2 times at 21 days intervals
  Interventions: Biological: LD Universal Influenza Vaccine Uniflu
- HD Universal Influenza Vaccine Uniflu (Active Comparator): high dose of Uniflu vaccine 0.5 ml (40 mkg of recombinant protein HBc-4M2eh) administrated intramuscularly 2 times at 21 days intervals
  Interventions: Biological: HD Universal Influenza Vaccine Uniflu
- Placebo (Placebo Comparator): saline 0.5 ml
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LD Universal Influenza Vaccine Uniflu — low dose Universal Influenza Vaccine Uniflu
  Arms: LD Universal Influenza Vaccine Uniflu
Biological: HD Universal Influenza Vaccine Uniflu — High dose Universal Influenza Vaccine Uniflu
  Arms: HD Universal Influenza Vaccine Uniflu
Biological: Placebo — Placebo saline
  Arms: Placebo

SUMMARY:
This is a single-site, randomized, double-blind, placebo-controlled study of Uniflu in fifty four (54) volunteers 18-60 years of age with a dose escalation.

All subjects will receive an intramuscular (IM) injection twice,with a 21 days interval between treatments.

DETAILED DESCRIPTION:
This is a single-site, randomized, double-blind, placebo-controlled study of Uniflu in fifty four (54) volunteers 18-60 years of age.

All subjects will receive an intramuscular (IM) injection twice,with a 21 days interval between treatments.

Subjects will undergo screening procedures within 6 days prior to first vaccination which will include medical history, vital signs, physical examination and safety blood and urine lab tests.

On the first treatment visit, eligible subjects will undergo pre-dose physical examination,vital signs, ECG, a blood sample will be drawn for circulating IgE. They receive an IM injection of either vaccine or placebo, according to the above treatment assignment, into the deltoid muscle. The subjects will remain under medical supervision for 72 hrs, after that time they will be released from the Clinical research center.

The second treatment will take place 21 days after the first vaccination. Procedures will be the same as on the first treatment visit.

Follow-up visits take place at 4th, 5th, 6th, 14th, 35th days. A Study Termination visit will take place at 42nd day of research. Adverse events (AEs) and changes in concomitant medications will be recorded, vital signs will be measured and the subjects will undergo physical examination and ECG. Blood and urine samples will be collected for safety.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 60 years old.
2. Healthy that verificated by vital signs, physical examination, blood and urine lab tests
3. Body mass index (BMI) from 18.5 to 30.5 weight >50 kg
4. Written informed consent.
5. Consent to the use of effective contraceptive methods throughout the study period.
6. Negative pregnancy test (for fertile women), consent to the use of effective contraceptive methods throughout the study period.

Exclusion criteria

1. Participation of a volunteer in any other study in the last 90 days; any vaccination in the last 30 days;
2. Vaccination within 6 months before the start of the study (including during participation in other clinical trials).
3. Symptoms of respiratory illness in the last 3 days.
4. Symptoms of any acute in the screening period.
5. Administration of immunoglobulins or other blood products for the last 3 months.
6. Taking immunosuppressive drugs and / or immunomodulators within 6 months before the start of the study.
7. Hypersensitivity or allergic reactions to the administration of any vaccine in medical history.
8. The presence of anaphylactic reactions, angioedema or other SAE to the administration of any vaccine in medical history.
9. Allergic reactions to vaccine components.
10. Seasonal allergy (at autumn period).
11. Acute or chronical desease or pathology from the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary and endocrine systems, which may influence the evaluation of the results of the study, in the anamnesis and also according to the screening examination data
12. Leukemia or any other blood disease or malignancy of other organs.
13. Thrombocytopenic purpura or bleeding disorders in medical history.
14. Seizures in medical history.
15. The presence or suspected presence of various immunosuppressive or immunodeficient state, including HIV infection.
16. Hepatitis B and C.
17. Tuberculosis.
18. Regular past or current use of narcotic drugs.
19. Pregnancy or breastfeeding.
20. Any conditions which may influence the evaluation of the results of the study, in the anamnesis and also according to the screening examination data.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2018-06-02 (Actual); Primary Completion 2018-12-02 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events in treatment vs control group | 42 days (from first visit to termination visit for each subject)
  Estimation the quantity of adverse events in treatment group vs control group

SECONDARY OUTCOMES:
Assessment of Immunogenicity | Time Frame: at days 1, 21, 42.
  Determination of antibody levels of IgG to M2e protein measured by IFA vs. baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Julia M Savateeva, PhD, Study Director — VA Pharma Limited Liability Company
Locations (1):
- Research Institute of Influenza, Saint Petersburg, Sankt-Peterburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided